CLINICAL TRIAL: NCT02058992
Title: Rozerem Tablets 8mg Drug Use Surveillance: Survey on Insomnia Associated With Sleep-onset Difficulty
Brief Title: Ramelteon Tablets 8mg Drug Use Surveillance: Survey on Insomnia Associated With Sleep-onset Difficulty
Status: Completed | Type: Observational
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Other Study IDs: 293-101; JapicCTI-132358 (Registry Identifier: JapicCTI); JapicCTI-R150751 (Registry Identifier: JapicCTI)
Record Dates: First submitted 2014-02-07; First posted 2014-02-11 (Estimated); Results first posted 2016-07-14 (Estimated); Last update posted 2016-07-14 (Estimated); Status verified 2016-06

CONDITIONS: Insomnia
Keywords: Drug therapy
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — ramelteon

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Ramelteon 8 mg administered orally once daily
  Interventions: Drug: Ramelteon

INTERVENTIONS:
Drug: Ramelteon — Ramelteon 8 mg tablets
  Other Names: Rozerem

SUMMARY:
The purpose of this study is to investigate the safety and efficacy of ramelteon (Rozerem) when used in the routine clinical setting in patients with sleep-onset difficulty associated with insomnia.

DETAILED DESCRIPTION:
This is a drug use surveillance planned to examine the safety and efficacy of ramelteon tablets when used in the routine clinical setting in patients with sleep-onset difficulty associated with insomnia (planned sample size, 3000)

The usual adult dosage is 8 mg of ramelteon administered orally once daily at bedtime.

ELIGIBILITY:
Inclusion Criteria:

1. Sleep-onset difficulty associated with insomnia

Exclusion Criteria:

1. Patients with previous history of hypersensitivity to an ingredient of Rozerem Tablets
2. Patients with severe liver dysfunction
3. Patients taking fluvoxamine maleate

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Insomnia
Sampling Method: Non-Probability Sample
Enrollment: 3339 (Actual)
Dates: Start 2010-07; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Postmarketing Group Manager, Study Chair — Takeda

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 557 investigative site in Japan from 30 July 2010 to 30 April 2013.
Pre-assignment Details: Participants with a historical diagnosis of insomnia who were facing difficulty in falling asleep in daily clinical practice were enrolled in single treatment group to receive ramelteon 8 milligram (mg).
Groups:
- Ramelteon: Ramelteon 8 mg, tablets, orally, once as daily clinical practice were observed for up to 4 weeks. A follow up of 2 weeks was carried out.
Period: Overall Study
Arm/Group | Ramelteon
Started | 3339
Completed | 3223
Not Completed | 116
Not completed — Lost to Follow-up | 4
Not completed — Protocol Violation | 92
Not completed — CRF Uncollected | 20

BASELINE CHARACTERISTICS:
Population: Safety analysis set was defined as participants who were enrolled and completed the study.
Arm/Group | Ramelteon
Number analyzed (Participants) | 3223
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.5 (18.9)
Age, Customized [Number; unit: participants]
  Less than (<) 65 years | 1379
  Greater than or equal to (>=)65 years to <75 years | 733
  >=75 years | 1111
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1935
  Male | 1288
Type of Sleep Disorder (Major Symptoms) [Number; unit: participants] — Sleep disorder was categorized on the basis of symptoms found in participants.
  participants
    Difficulty falling asleep | 1966
    Difficulty getting sound sleep | 302
    Difficulty staying asleep | 458
    Early morning awakening | 50
    Unknown | 447
Degree of Sleep Disorder [Number; unit: participants] — Degree of sleep disorder of participants were categorized on the basis of the judgement of the investigator as mild, moderate and severe.
  participants
    Mild | 1354
    Moderate | 1569
    Severe | 300
Duration of Insomnia [Mean (Standard Deviation); unit: years] | 1.13 (2.45)
Duration of Insomnia [Number; unit: participants]
  < 1 year | 1522
  >=1 year to <3 years | 241
  >=3 to < 5 years | 107
  >=5 years | 135
  Unknown | 1218
Presence of Complications [Number; unit: participants]
  Had Complications | 2618
  Had No Complications | 605
Breakdown of complications [Number; unit: participants] — Participants could be counted in more than 1 category (including duplicates).
  participants
    Hypertension | 1206
    Dyslipidaemia | 694
    Mental disease | 495
    Diabetes mellitus | 419
    Heart or cerebrovascular disease | 393
    Renal and urinary disorders | 158
    Hepatobiliary disorders | 133

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Reporting One or More Adverse Drug Reactions
Description: Adverse drug reactions are defined as adverse events (AE) which are in the investigator's opinion of causal relationship to the study treatment. AE are defined as any unfavorable and unintended signs, symptoms or diseases temporally associated with the use of a medicinal product reported from the first dose of study drug to the last dose of study drug.
Time Frame: Baseline up to 6 weeks
Population: Safety analysis set was defined as participants who were enrolled and completed the study.
Measure: Number; unit: participants
Arm/Group | Ramelteon
Number analyzed (Participants) | 3223
participants | 109

2. Primary Outcome: Number of Participants Reporting One or More Serious Adverse Drug Reactions
Description: Serious adverse drug reactions are defined as serious adverse events (SAE) which are in the investigator's opinion of causal relationship to the study treatment. An SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly.
Time Frame: Baseline up to 6 weeks
Population: SAS was defined as participants who were enrolled and completed the study.
Measure: Number; unit: participants
Arm/Group | Ramelteon
Number analyzed (Participants) | 3223
participants | 1

3. Secondary Outcome: Sleep Status: Sleep Onset Latency
Description: Sleep status was determined by measuring the sleep onset latency, defined as the length of time taken from lying down for the night until sleep onset.
Time Frame: Baseline and Week 4
Population: The efficacy assessment population was defined as participants whose efficacy data at baseline and at least 1 post-baseline time points was available.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Ramelteon
Number analyzed (Participants) | 1429
minutes
  Baseline | 89.8 (66.7)
  Week 4 | 47.1 (46.2)

4. Secondary Outcome: Sleep Status: Total Sleep Time
Description: Sleep status was determined by measuring the total sleep time, defined as the amount of actual sleep time during a sleep episode.
Time Frame: Baseline and Week 4
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Ramelteon
Number analyzed (Participants) | 1292
hours
  Baseline | 6.49 (2.00)
  Week 4 | 7.31 (1.72)

5. Secondary Outcome: Sleep Status: Number of Awakenings
Description: Sleep status of participants was assessed and summarized by calculating the number of times participants had awaken from the time of start of the investigation.
Time Frame: Baseline and Week 4
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: number of awakenings
Arm/Group | Ramelteon
Number analyzed (Participants) | 1401
number of awakenings
  Baseline | 2.1 (1.6)
  Week 4 | 1.2 (1.2)

6. Secondary Outcome: Percentage of Participants Who Responded With Improvement on the Patient Global Impression (PGI) Scale at Week 4
Description: PGI is a participant rated instrument to measure participant's change in overall status on a 7-point scale. 7 items on scale include sleep onset, sleep time, sleep quality, morning awakening, morning tiredness, daytime somnolence, and daytime physical condition/function. Participants provide their response on a PGI questionnaire. The results of survey using the PGI questionnaire was scored, summarized and assessed. Total score range from 1 (very much improved) to 7 (very much worse). Percentage of participants with improvement rated as "much better" or "a little better" were reported for sleep onset,time, quality; morning awakening, tiredness and daytime sleepiness, physical condition.
Time Frame: Week 4
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Ramelteon
Number analyzed (Participants) | 2788
percentage of participants
  Sleep onset | 69.6
  Sleep time | 63.8
  Sleep quality | 64.8
  Morning awakening | 54.0
  Morning tiredness | 52.9
  Daytime sleepiness | 51.9
  Daytime physical condition/function | 55.8

ADVERSE EVENTS:
Time Frame: Baseline up to 6 weeks
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment. Only adverse drug reactions were collected in this study.
Arm/Group | Ramelteon
Serious Adverse Events (participants affected / at risk) | 1/3223
Other Adverse Events (participants affected / at risk) | 37/3223
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ramelteon (N=3223)
Death (General disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ramelteon (N=3223)
Somnolence (Nervous system disorders) | 37

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi-site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.